CLINICAL TRIAL: NCT04752267
Title: Novel Dynamic PET Kinetics and MRI Radiomics Analyses in Brain Tumors
Brief Title: 18F-FMAU PET/CT and MRI for the Detection of Brain Tumors in Patients With Brain Cancer or Brain Metastases
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6B-20-1; NCI-2021-00706 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 6B-20-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Glioma; Malignant Brain Neoplasm; Metastatic Breast Carcinoma; Metastatic Colon Carcinoma; Metastatic Kidney Carcinoma; Metastatic Lung Carcinoma; Metastatic Malignant Neoplasm in the Brain; Metastatic Melanoma; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Stage IV Colon Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Stage IVA Colon Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Colon Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Stage IVC Colon Cancer AJCC v8
MeSH Terms: conditions — Glioma; Brain Neoplasms; Breast Neoplasms; Colonic Neoplasms; Carcinoma, Renal Cell; Lung Neoplasms; Melanoma | interventions — clevudine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (18F-FMAU, PET/CT, mpMRI) (Experimental): Patients receive 18F-FMAU intravenously (IV) and undergo a PET/CT scan over 60 minutes. Patients then undergo standard of care mpMRI over approximately 45 minutes.
  Interventions: Procedure: Computed Tomography; Drug: 18F-FMAU; Procedure: Multiparametric Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: 18F-FMAU — Given IV
  Other Names: Fluorine F 18 d-FMAU
Procedure: Multiparametric Magnetic Resonance Imaging — Undergo mpMRI
  Other Names: MP-MRI; mpMRI; Multi-parametric MRI; Multiparametric MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This early phase I trial tests the use of a radioactive tracer (a drug that is visible during an imaging test) known as 18F-FMAU, for imaging with positron emission tomography/computed tomography (PET/CT) in patients with brain cancer or cancer that has spread to the brain (brain metastases). A PET/CT scan is an imaging test that uses a small amount of radioactive tracer (given through the vein) to take detailed pictures of areas inside the body where the tracer is taken up. 18F-FMAU may also help find the cancer and how far the disease has spread. Magnetic resonance imaging (MRI) is a type of imaging test used to diagnose brain tumors. 18F-FMAU PET/CT in addition to MRI may make the finding and diagnosing of brain tumor easier.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the correlation between multiparametric magnetic resonance imaging (mpMRI) radiomics and dynamic 2'-fluoro-5-methyl-1-beta-D-arabinofuranosyluracil (FMAU) PET kinetic analysis parameters.

II. Explore the different pattern in radiomics mpMRI and FMAU PET kinetic analysis parameters between patients with presence or absence of recurrent tumor.

OUTLINE:

Patients receive 18F-FMAU intravenously (IV) and undergo a PET/CT scan over 60 minutes. Patients then undergo standard of care mpMRI over approximately 45 minutes.

After completion of study intervention, patients are followed up at 24-96 hours after their 18F-FMAU PET/CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, both men and women
* Documented history of either primary brain tumor (e.g. glioma) or metastatic brain tumor from another primary cancer (e.g. lung, breast, colon, melanoma, kidney)
* Documented radiation therapy regardless of treatments prior to radiation therapy

Exclusion Criteria:

* Unable to give consent
* Inability to remain motionless during imaging studies
* Intractable seizures
* Claustrophobia
* Implantable devices incompatible with magnetic resonance (MR) environment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Correlation between multiparametric magnetic resonance imaging (mpMRI) radiomics and dynamic fluorine F 18 (18F)-FAMU (FMAU) positron emission tomography (PET) kinetic analysis parameters | Up to 1 year
  Scatter plots will be used to illustrate the pattern of correlation. For normality distributed data, Pearson correlation will be used; otherwise, Spearman correlation will be used. There will be 90 pairs of correlations. To further confirm the robustness of the correlation finding, the Benjamini-Hochberg procedure will be applied to prevent false discovery.
Different pattern in radiomics mpMRI and FMAU PET kinetic analysis parameters | Up to 1 year
  Interesting patterns will be observed at individual subject level for the difference between presence or absence of recurrent tumor, which defined as either underlying immunohistochemistry (Ki67-MIB proliferation marker, when tissue sample is available, or a binary proxy marker of subsequent clinical management decision (with wait-and-watch strategy for 1 month after imaging studies considered as "absence" of recurrent tumor, otherwise marked as "presence" of recurrent tumor). Heatmap will be used with subject identification as x-axis and each radiomic/kinetic feature as y-axis. Features will be divided by categories to facilitate the visualization of patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Jadvar, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States